CLINICAL TRIAL: NCT01793116
Title: Time Limited Observational Study of the Moderately Preterm Infant (29 0/7 - 33 6/7 Weeks)
Brief Title: Generic Database of Moderate Preterm Infants
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0049; U10HD021364 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD021373 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD040461 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Moderate Preterm
Keywords: NICHD Neonatal Research Network; Moderately Preterm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 11 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry of moderate preterm infants, born alive at 29-33 weeks gestational age, in NICHD Neonatal Research Network (NRN) centers. The registry collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The information collected is not specific to a disease or treatment (i.e., it is "generic"). Data are analyzed to find associations and trends between baseline information, treatments, and infant outcome, and to develop future NRN trials.

DETAILED DESCRIPTION:
The Moderate Preterm Registry is a registry of moderate preterm infants (29-33 weeks gestational age) born alive in NICHD Neonatal Research Network (NRN) centers. The purpose is to collect baseline and outcome data in a uniform manner on a cohort of infants.

The registry collects observational baseline data on both mothers and infants, and the therapies used and outcomes of the infants. The information collected is not specific to a disease or treatment (i.e., it is "generic"). Baseline data is collected soon after admission to the NICU; outcome data is collected at the time of death or discharge from the hospital. The data collected includes information on:

* Demographics of mother and infant
* Mother's health (e.g., pregnancy history and complications)
* Labor and deliver (e.g., rupture of the membranes, steroids and antibiotics given, mode of delivery)
* Infant's health (gestational age, Apgar scores, weight, length, delivery room resuscitation, respiratory support, etc.)
* Infant's medical outcome (heart, lung, nervous system, gastrointestinal system, hearing, and vision, known infections, and major malformations/syndromes, and mortality or number of days hospitalized).

These data are used: to examine associations between baseline characteristics, treatments, and outcomes; to track trends in incidences of disease and effectiveness of therapies; and to identify questions requiring additional in-depth research.

Informed Consent: As required by local IRBs.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 29-33 weeks
* Inborn infants and outborn infants admitted by 72 hours.

Exclusion Criteria:

* None

Ages: 29 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Moderately preterm infants born at 29 0/7 weeks to 33 6/7 weeks-both inborn and outborn but admitted prior to 72 hours at NRN centers will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 7057 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of infants born moderately preterm | up to 2 years
  Number of infants born between 29-33 weeks gestational age at 18 participating NRN centers.

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C Walsh, MD, MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N Goldberg, MD, Principal Investigator — Duke University; Barbara J Stoll, MD, Principal Investigator — Emory University; Brenda B Poindexter, MD, MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingha; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Seetha Shankaran, MD, Principal Investigator — Wayne State University; William Truog, MD, Principal Investigator — Abbot R Laptook, MD Study Principal Investigator Brown University, Women & Infants Hospital of Rhode Island Michele C Walsh, MD MS Study Principal Investigator Case Western Reserve University, Rainbow Babies and Children's Hospital Ronald N Goldberg,; Barbara Schmidt, MD, MSc, Principal Investigator — University of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Leif Nelin, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — http://www.nichd.nih.gov/about/org/der/branches/ppb/pages/overview.aspx